CLINICAL TRIAL: NCT00075231
Title: A Randomized, Open-Label Study Exploring a Simplified Kaletra® (Lopinavir/Ritonavir)-Based Therapy Versus a Sustiva® (Efavirenz)-Based Standard of Care in Previously Non-Treated HIV-Infected Subjects
Brief Title: A Simplified Kaletra® (Lopinavir/Ritonavir)-Based Therapy Versus a Sustiva® (Efavirenz)-Based Standard of Care in Previously Non-Treated HIV-Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M03-613
Record Dates: First submitted 2004-01-06; First posted 2004-01-08 (Estimated); Last update posted 2006-10-02 (Estimated); Status verified 2006-09

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir; lamivudine, zidovudine drug combination; Lamivudine; Zidovudine; efavirenz

INTERVENTIONS:
Drug: Kaletra® (lopinavir/ritonavir)
Drug: Combivir® (lamivudine, zidovudine)
Drug: Sustiva® (efavirenz)

SUMMARY:
The purpose of this study is to determine whether a simplified lopinavir-ritonavir based therapy will continue to keep the viral load to very low levels after initial treatment with a combination of Kaletra® (lopinavir/ritonavir) plus Combivir® (lamivudine/zidovudine).

ELIGIBILITY:
Inclusion Criteria

* Subject is at least 18 years of age.
* Subject is confirmed HIV positive and in the investigator's opinion requires antiretroviral (ARV) therapy.
* Subject is naïve to HIV ARV therapy or has received < 7 days total of any HIV ARV therapy > 30 days prior to study drug administration.
* Subject's HIV RNA is >= 1000 copies/mL at screening.
* If sexually active, subject agrees to use safe sex practices to reduce risk of HIV transmission (e.g., male or female condom, vaginal dam, etc.).
* If female, the results of a urine pregnancy test performed at screening and on Day 1/Baseline are both negative.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:

  * A. Condoms, sponge, foams, jellies, diaphragm or intrauterine device.
  * B. A vasectomized partner.
  * C. Total abstinence from sexual intercourse.
* Subject is not breastfeeding.
* Subject's vital signs, physical examination, and laboratory results do not exhibit evidence of acute illness.
* Subject has a Karnofsky score greater than or equal to 70.
* Subject agrees not to take any drugs during the study, including over-the-counter medicines, vitamins, mineral supplements, herbal preparations, alcohol, or recreational drugs without the knowledge and permission of the investigator.
* Subject has not been treated for an active AIDS-defining opportunistic infection within 30 days of initiating study drug.
* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

Exclusion Criteria

* A subject will be excluded from the study if he/she meets any of the following criteria:
* Subject has a history of an allergic reaction or significant sensitivity to lopinavir, ritonavir, lamivudine, zidovudine, efavirenz, or to any inert materials contained in the study drug formulations.
* Subject has significant history of cardiac, renal, neurologic, psychiatric, oncologic, endocrinologic, metabolic, or hepatic disease that would, in the opinion of the investigator, adversely affect his/her participation in this study.
* Subject is currently taking any drug (medicinal or herbal) that is contraindicated and/or not to be co-administered with any of the three study drugs as defined in the current locally approved prescribing information.
* Subject has a history of drug and/or alcohol abuse or psychiatric illness that in the investigator's opinion could preclude compliance with the protocol.
* Subject is receiving immunomodulatory agents, colony stimulating factor, bone marrow stimulants (e.g., erythropoietin [Procrit®, Epogen®] or filgrastim [Neupogen®]), ganciclovir, interferon-alpha, and other bone marrow suppressive or cytotoxic agents.
* The TRUGENE HIV-1 resistance report indicates resistance or possible resistance to the study reverse transcriptase inhibitor(s) [RTI(s)] (efavirenz, lamivudine or zidovudine) OR the presence of any mutation in the protease gene leading to an amino acid substitution at the following loci: 8, 30, 32, 46, 47, 48, 50, 54, 82, 84, or 90 OR four or more mutations at the following loci: 10, 20, 24, 36, 53, 63, or 71.
* Screening laboratory analyses show any of the following abnormal laboratory results: Presence of Hepatitis B surface antigen (HBsAg); Hemoglobin <= 9.5 g/dL; Absolute neutrophil count <= 1000 cells/mL; Platelet count <= 50,000 per mL; ALT (SGPT) or AST (SGOT) >= 3.0 x Upper Limit of Normal (ULN); Fasting Triglycerides > 750 mg/dL; Fasting Cholesterol > 300 mg/dL; Creatinine >= 1.5 x Upper Limit of Normal (ULN); Fasting serum glucose > 126 mg/dL
* Subject is taking a prescribed lipid lowering medication such as HMG-CoA Reductase Inhibitors (statin) or fibrate medications.
* Subject has a history of diabetes mellitus.
* Subject has received any investigational drug or vaccine within 30 days prior to study drug administration.
* For any reason, subject is considered by the investigator to be an unsuitable candidate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-12

PRIMARY OUTCOMES:
Proportion of subjects with a plasma HIV RNA level below 50 copies/mL at Week 96.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara da Silva, M.D., Study Director — Abbott
Locations (1):
- Fountain Valley Regional Hospital and Medical Center, Fountain Valley, California, United States

REFERENCES:
- [Derived] Brown TT, McComsey GA, King MS, Qaqish RB, Bernstein BM, da Silva BA. Loss of bone mineral density after antiretroviral therapy initiation, independent of antiretroviral regimen. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):554-61. doi: 10.1097/QAI.0b013e3181adce44. PMID 19512937
- [Derived] Cameron DW, da Silva BA, Arribas JR, Myers RA, Bellos NC, Gilmore N, King MS, Bernstein BM, Brun SC, Hanna GJ. A 96-week comparison of lopinavir-ritonavir combination therapy followed by lopinavir-ritonavir monotherapy versus efavirenz combination therapy. J Infect Dis. 2008 Jul 15;198(2):234-40. doi: 10.1086/589622. PMID 18540803